CLINICAL TRIAL: NCT07086118
Title: Efficacy of Dexamethasone Versus Metoclopramide for Prophylaxis of Nausea and Vomiting After Cataract Surgery: A Double-blind Randomized Controlled Study
Brief Title: Dexamethasone Versus Metoclopramide for Prophylaxis of Nausea and Vomiting After Cataract Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, sarah mohamed, lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 0307296
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Cataract; Dexamethasone
Keywords: dexamethasone; cataract surgery
MeSH Terms: conditions — Cataract | interventions — Saline Solution; Metoclopramide; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group p (Placebo Comparator): patients will receive 0.9% normal saline
  Interventions: Other: 0.9% normal saline
- group M (Active Comparator): patients will receive 10 mg metoclopramide
  Interventions: Drug: Metoclopramide 10mg
- group D (Active Comparator): patients will receive 8 mg dexamethasone
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Other: 0.9% normal saline — patients in group P will receive 0.9% normal saline
  Other Names: group P
  Arms: group p
Drug: Metoclopramide 10mg — patients in group M will receive 10 mg metoclopramide
  Other Names: group M
  Arms: group M
Drug: Dexamethasone — patients in group D will receive 8 mg dexamethasone
  Other Names: group D
  Arms: group D

SUMMARY:
Postoperative nausea and vomiting (PONV) is a common consequence of ambulatory surgery, affecting up to 80% of high-risk patients and 20-30% overall. Despite being widespread, a prior survey found that patients are more averse to PONV than pain and other significant postoperative problems. Furthermore, even mild cases of PONV can have serious repercussions, such as postanesthesia care unit (PACU) workflow disruption, delayed discharges, higher medical costs, and lower patient satisfaction.PONV following intraocular surgery can be unpleasant and may lead to serious complications including suprachoroidal hemorrhage (SCH). SCH is a potentially serious condition that occurs when the posterior ciliary arteries or vortex veins burst, resulting in blood in the suprachoroidal region.

The hypothesis is that dexamethasone will lower the incidence of PONV after cataract surgery when compared with metoclopramide.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a common consequence of ambulatory surgery, affecting up to 80% of high-risk patients and 20-30% overall.(1) Despite being widespread, a prior survey found that patients are more averse to PONV than pain and other significant postoperative problems.(2) Furthermore, even mild cases of PONV can have serious repercussions, such as postanesthesia care unit (PACU) workflow disruption, delayed discharges, higher medical costs, and lower patient satisfaction.(3)PONV following intraocular surgery can be unpleasant and may lead to serious complications including suprachoroidal hemorrhage (SCH).(4) SCH is a potentially serious condition that occurs when the posterior ciliary arteries or vortex veins burst, resulting in blood in the suprachoroidal region.(5)

Several medications are proved to be effective for prevention of nausea and vomiting like steroids, dopamine antagonists and serotonin antagonists. PONV is best prevented and treated with selective serotonin receptor antagonists. Although serotonin receptor antagonists are more successful than metoclopramide and dexamethasone in preventing and treating PONV, their usage is restricted due to their expensive cost and limited availability in resource-poor facilities.(6) In an attempt to decrease the incidence of PONV in the ambulatory setting, several anti-emetics have been studied.(7) For decades, metoclopramide has been a popular antiemetic due to its dose-dependent activity on central dopaminergic D2 receptors, central and peripheral 5-HT3 receptors, and peripheral 5-HT4 receptors. Despite inconsistent results, it is nevertheless commonly used in clinical practice to prevent nausea and vomiting after surgery.(8) Dexamethasone was utilized as a standalone medication during surgery for both pediatric and adult patients.(9) Recently, there has been a suggestion that dexamethasone, which has been shown to be more effective in preventing nausea and is thought to lower 5-HT levels in the central nervous system, could lower the incidence of PONV.(10)

The hypothesis is that dexamethasone will lower the incidence of PONV after cataract surgery when compared with metoclopramide.

Aim of the work:

The present study aims to test the efficacy of dexamethasone and metoclopramide in prevention of PONV in patients undergoing cataract surgery.

Primary outcome:

• Incidence of PONV

Secondary outcomes:

* Number of patients took antiemetic drug in 24h
* Postoperative pain score

Patients :

Study settings:

This study will be conducted in ophthalmology department, Alexandria university hospitals.

Study design:

Placebo-controlled, double blind, randomized, prospective study

Sample size calculation:

Study population:

All patients will be randomized 1:1 using a sealed envelope method. Patients will be divided into three equal groups:

Group P: patients will receive 0.9% normal saline

Group M: patients will receive 10 mg metoclopramide Group D: patients will receive 8 mg dexamethasone

Methods:

Preoperative evaluation and preparation:

During preoperative visit, evaluation of patients will be carried out through proper history taking, clinical examination and routine laboratory investigations including complete blood picture, coagulation profile, blood urea, serum creatinine, serum electrolytes and any other investigation needed.

Pre-anesthetic preparation and premedication:

* Informed written consent, from all individual participants who will be included in this study will be taken during preoperative visit.
* Patients should be trained during preoperative visit on a visual analogue scale (VAS), with 0 corresponding to no pain and 10 to the worst pain imaginable

On arrival to operative theatre, intravenous cannula will be inserted and standard monitoring will be established using multichannel monitor (Carescape Monitor B650, GE Healthcare Finland) to monitor the following in both groups:

* Electrocardiogram (ECG) for heart rate and rhythm. (Beats/min).
* Non-invasive measurement of arterial blood pressure. (Mean blood pressure in mmHg).
* Pulse oxygen saturation. (SpO2%). Before sedation, patients will be randomly allocated to receive one of three drugs. Three 2-mL syringes containing either 8 mg dexamethasone,10 mg metoclopramide, or 0.9% saline per syringe will be prepared by an anesthetist who is not one of the observers. Syringes will be marked with a coded label. Patients in group P will receive 0.9% normal saline, group M will receive 10 mg metoclopramide and group D will receive 8 mg dexamethasone before sedation. All patients will be sedated with 0.025 mg /kg midazolam, 0.25 mg/kg ketamine and 0.05 mg/kg nalbuphine. Peribulbar block with 2 ml lidocaine 2% and 3 ml bupivacaine 0.5% will be given to all patients.

The rescue antiemetic will be ondansetron 4 mg IV, which will be given for prolonged nausea (exceeding 10 min) or vomiting or at the patient's request and will be repeated if necessary. Pain will be assessed using VAS. Nausea will be assessed using a linear numerical scale of 0-3 (0=none, 1=mild, 2=moderate, 3=severe). The rescue analgesic will be intravenous ketorolac 30 mg if VAS >3. Nausea refers to the unpleasant sensation of wanting to vomit, while vomiting is the forceful ejection of gastric contents from the mouth.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-80 years, both sexes.
* ASA physical status class I to III.

Exclusion Criteria:

* history of motion sickness
* patients with gastrointestinal disorders or gastro-oesophageal reflux
* patients taking medications with known antiemetic activity
* previous postoperative vomiting
* allergy to bupivacaine
* allergy to metoclopramide or dexamethasone

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
number of patients with nausea and vomiting | postoperative day 1
  number

SECONDARY OUTCOMES:
vas score | postoperative day 1
  score
number of patients requiring antiemetic | postoperative day1
  number
incidence of dizziess, pruritis and headache | postoperative day 1
  number

CONTACTS AND LOCATIONS:
Overall Officials: sarah m elgamal, MD, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bilgin TE, Birbicer H, Ozer Z, Doruk N, Tok E, Oral U. A comparative study of the antiemetic efficacy of dexamethasone, ondansetron, and metoclopramide in patients undergoing gynecological surgery. Med Sci Monit. 2010 Jul;16(7):CR336-41. PMID 20581776